CLINICAL TRIAL: NCT01986907
Title: A 12 Months, Prospective, Multicenter, Open-label, Single Arm Interventional Study Assessing the Safety and Tolerability of 0.5 mg Ranibizumab in Mono/Bilateral Wet AMD Patients in Eyes With (Best-Corrected Distance Visual Acuity) BCVA Below 2/10 and/or Second Affected Eye
Brief Title: Safety and Tolerability of Ranibizumab in Mono/Bilateral Wet Age Related Macular Degeneration (w-AMD) Patients in Eyes With BCVA<2/10 and/or 2nd Affected Eye
Acronym: TWEYES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002AIT02; 2013-003333-15 (EudraCT Number)
Record Dates: First submitted 2013-11-12; First posted 2013-11-19 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-05

CONDITIONS: Wet Age Related Macular Degeneration
Keywords: wet AMD; macular degeneration; ranibizumab; mono-bilateral; poor visual acuity; retinal disease; eye disease; Angiogenesis Inhibitors; Angiogenesis Modulating Agents
MeSH Terms: conditions — Macular Degeneration; Retinal Diseases; Eye Diseases | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ranibizumab (Experimental): Administered as an Intravitreal injection
  Interventions: Drug: ranibizumab

INTERVENTIONS:
Drug: ranibizumab — All patients will receive ranibizumab 0.5 mg/0.05 ml according to approved label: treatment is given monthly until maximum VA is achieved (i.e. stable VA for three consecutive monthly assessments performed while on ranibizumab treatment). Thereafter according to approved label, patients should be monitored monthly for visual acuity and treatment is to be resumed when monitoring indicates loss of visual acuity due to disease activity. Monthly injections should then be administered until stable visual acuity is reached again for three consecutive monthly assessments (implying a minimum of two injections).

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ranibizumab in patients affected by wet age related macular degeneration (wAMD).

ELIGIBILITY:
Inclusion Criteria

Male or female patients aged 50 years or above Willing and capable to provide informed written consent Eye(s) eligible for ranibizumab treatment, with a BCVA below 2/10 due to wet AMD and/or Second eye eligible for ranibizumab treatment, with first eye treated (currently or previously) with ranibizumab, whichever BCVA. In bilateral wAMD patients, the second eye can be included only if the first eye has been treated at least 14 days before with ranibizumab

Exclusion Criteria:

Active intraocular inflammation (grade trace or above) in either eye Any ocular or periocular active infection (current or suspected), e.g. conjunctivitis, keratitis, scleritis, uveitis, endophtalmitis, in either eye Risk factors for retinal pigment epithelial tear (including pigment epithelial retinal detachment) Ocular disorders that may confound interpretation of results compromise visual acuity or require medical or surgical intervention during the study period including cataract, retinal vascular occlusion, retinal detachment or macular hole Uncontrolled glaucoma in either eye (IOP ≥ 30 mmHg on medication or according to investigator's judgment) History of vitrectomy in the study eye History of stroke or transient ischemic attack Systemic treatment with any VEGF inhibitor in the 90 days prior to study enrollment Ocular treatment of the study eye with any anti-angiogenic drugs within 1 month prior to study enrollment Any intraocular surgery in the study eye within 28 days prior to enrollment Women of childbearing potential UNLESS using effective contraception during treatment Pregnant or lactating women Simultaneous participation in a study that includes administration of any investigational drug Known hypersensitivity to ranibizumab or any component of the ranibizumab formulation Inability to comply with study procedures.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1049 (Actual)
Dates: Start 2014-03-04 (Actual); Primary Completion 2016-06-15 (Actual); Study Completion 2016-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (84):
- Italy (84):
  - Novartis Investigative Site, Alessandria, AL
  - Novartis Investigative Site, Casale Monferrato, AL
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Acquaviva delle Fonti, BA
  - Novartis Investigative Site, Putignano, BA
  - Novartis Investigative Site, Terlizzi, BA
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Belluno, BL
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Desenzano del Garda, BS
  - Novartis Investigative Site, Bolzano, BZ
  - Novartis Investigative Site, Cagliari, CA
  - Novartis Investigative Site, Larino, CB
  - Novartis Investigative Site, Caserta, CE
  - Novartis Investigative Site, Chieti, CH
  - Novartis Investigative Site, Ceva, CN
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Como, CO
  - Novartis Investigative Site, San Feramo Della Battaglia, CO
  - Novartis Investigative Site, Acireale, CT
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Catanzaro, CZ
  - Novartis Investigative Site, Forlì, FC
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Rapallo, GE
  - Novartis Investigative Site, Crotone, KR
  - Novartis Investigative Site, Tricase, LE
  - Novartis Investigative Site, Terracina, LT
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milazzo, ME
  - Novartis Investigative Site, Cinisello Balsamo, MI
  - Novartis Investigative Site, Legnano, MI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Vizzolo Predabissi, MI
  - Novartis Investigative Site, Nuoro, NU
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Piacenza, PC
  - Novartis Investigative Site, Camposampiero, PD
  - Novartis Investigative Site, Monselice, PD
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Città di Castello, PG
  - Novartis Investigative Site, Foligno, PG
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Pordenone, PN
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Correggio, RE
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Civitavecchia, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Riccione, RN
  - Novartis Investigative Site, Eboli, SA
  - Novartis Investigative Site, Salerno, SA
  - Novartis Investigative Site, Sondrio, SO
  - Novartis Investigative Site, Sarzana, SP
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Savona, SV
  - Novartis Investigative Site, Taranto, TA
  - Novartis Investigative Site, Teramo, TE
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Terni, TR
  - Novartis Investigative Site, Trieste, TS
  - Novartis Investigative Site, Conegliano, TV
  - Novartis Investigative Site, Treviso, TV
  - Novartis Investigative Site, Udine, UD
  - Novartis Investigative Site, Busto Arsizio, VA
  - Novartis Investigative Site, Somma Lombardo, VA
  - Novartis Investigative Site, Varese, VA
  - Novartis Investigative Site, Santorso, VI
  - Novartis Investigative Site, Vicenza, VI
  - Novartis Investigative Site, Legnago, VR
  - Novartis Investigative Site, Negrar, VR
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Borgomanero
  - Novartis Investigative Site, Galliate
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Pozzuoli

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from investigative sites located in Italy.
Pre-assignment Details: This reporting group includes all treated patients (one eye or both eyes)
Groups:
- Ranibizumab: patients treated with 0.5mg ranibizumab
Period: Overall Study
Arm/Group | Ranibizumab
Started (All treated participants (one eye or both eyes) (Safety Analysis Set)) | 936
Completed | 774
Not Completed | 162
Not completed — Adverse Event | 11
Not completed — Unsatisfactory therapeutic effect | 24
Not completed — Protocol Violation | 4
Not completed — Withdrawal by Subject | 76
Not completed — Lost to Follow-up | 38
Not completed — Death | 9

BASELINE CHARACTERISTICS:
Population: All treated participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 936
Age, Continuous [Mean (Standard Deviation); unit: years] | 78.68 (7.34)
Age, Customized [Count of Participants; unit: Participants]
  18 to less than 65 years | 33
  65 to 74 years | 212
  75 to 84 years | 483
  85 years and older | 208
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 582
  Male | 354
Treatment by Eye [Count of Participants; unit: Participants] — Unilateral (one eye) or Bilateral (both eyes) treated
  Participants
    Unilateral treatment | 823
    Bilateral treatment | 113

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Systemic Drug-related Adverse Events
Description: Monitoring and recording all adverse events, including serious adverse events.
Time Frame: Baseline to Month 12
Population: Safety Set
Measure: Number; unit: participants
Arm/Group | Ranibizumab
Number analyzed (Participants) | 936
participants
  Serious Adverse Event | 3
  Non Serious Adverse Event | 0

2. Secondary Outcome: Overall Number of Ranibizumab Injections
Time Frame: Baseline to month 12
Population: Safety Set
Measure: Mean (Standard Deviation); unit: injections per patient
Arm/Group | Ranibizumab
Number analyzed (Participants) | 936
injections per patient | 5.97 (3.62)

3. Secondary Outcome: Time Interval Between Injections in Bilateral Disease
Description: Mean number of days between two consecutive injections per eye
Time Frame: Baseline to month 12
Population: This analysis population includes all eyes naïve to ranibizumab, i.e., had not been treated with the study medication (or with the equivalent commercial formulation) before the first study drug injection, regardless of whether the contralateral eye had been treated.
Measure: Mean (Standard Deviation); unit: days
Units Other Than Participants: eyes
Arm/Group | Ranibizumab
Number analyzed (Participants) | 936
Number analyzed (eyes) | 771
days | 51.94 (26.56)

4. Secondary Outcome: Mean Number of Injections Per Patient
Description: Number of injections per patient
Time Frame: Baseline to month 12
Population: Safety set
Measure: Mean (Standard Deviation); unit: injections
Groups:
- Ranibizumab Overall: patients treated with 0.5mg ranibizumab
Arm/Group | Ranibizumab Overall | Unilaterally Treted | Bilaterally Treated
Number analyzed (Participants) | 936 | 823 | 113
injections | 5.97 (3.62) | 5.35 (2.88) | 10.55 (4.98)

5. Primary Outcome: Number of Eyes With Ocular Drug-related Adverse Events
Description: Monitoring and recording all adverse events, including serious adverse events.
Time Frame: Baseline to Month 12
Population: Safety Set
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Ranibizumab
Number analyzed (Participants) | 936
Number analyzed (eyes) | 1049
eyes
  Serious Adverse Event | 1
  Non Serious Adverse Event | 8

ADVERSE EVENTS:
Time Frame: Adverse events are reported from time of first treatment until study exit (approximately 12 months)
Description: This reporting group (Safety Population) includes all treated participants (one or both eyes).
Groups:
- Ranibizumab 0.5 mg: Ranibizumab 0.5 mg
Arm/Group | Ranibizumab 0.5 mg
All-Cause Mortality (participants affected / at risk) | 9/936
Serious Adverse Events (participants affected / at risk) | 63/936
Other Adverse Events (participants affected / at risk) | 76/936
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=936)
Anaemia (Blood and lymphatic system disorders) | 2
Bone marrow disorder (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrioventricular block (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 3
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Goitre (Endocrine disorders) | 1
Ocular hypertension (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vitreous haemorrhage (Eye disorders) | 1
Faecaloma (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Large intestine polyp (Gastrointestinal disorders) | 1
Lumbar hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
General physical health deterioration (General disorders) | 1
Hepatic lesion (Hepatobiliary disorders) | 1
Escherichia sepsis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Pyelonephritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 7
Humerus fracture (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Pancreatic injury (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 1
Myasthenia gravis (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 3
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Mastectomy (Surgical and medical procedures) | 1
Transurethral prostatectomy (Surgical and medical procedures) | 1
Peripheral artery stenosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=936)
Cataract (Eye disorders) | 10
Conjunctival haemorrhage (Eye disorders) | 13
Neovascular age-related macular degeneration (Eye disorders) | 34
Pyrexia (General disorders) | 10
Influenza (Infections and infestations) | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.